CLINICAL TRIAL: NCT00997061
Title: SCOT Registry: Small Cell Lung Cancer Treatment and Outcome
Acronym: SCOT
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112791
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Lung Cancer, Small Cell
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HYCAMTIN
  Interventions: Drug: HYCAMTIN

INTERVENTIONS:
Drug: HYCAMTIN — Observing patients on HYCAMTIN and other drugs for SCLC.

SUMMARY:
The registry is an international, multicenter, observational registry of newly diagnosed patients with SCLC.

Data will be entered into an electronic CRF (eCRF) via Internet access. Treatment plan remains the responsibility of the patient's physician and data collected in this registry will reflect a "real world" approach of the diagnosis and treatment of patients with SCLC.

Approximately 60 centres in 13 countries will take part in this registry. It is expected that about 500 patients will be recruited during a period of 6 to 9 months according to the feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female >/= 18 years
* Diagnosis of small cell lung cancer
* Patient newly diagnosed with SCLC
* Has given written informed consent (if applicable)

Exclusion Criteria:

* Concurrent history of other neoplasm, except curatively treated basal cell skin cancer or adequately treated in-situ carcinoma of the cervix.
* Patient presenting with recurrence of SCLC.
* Patients who has received any chemotherapy for the SCLC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly Diagnosed SCLC patients
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2009-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Registry with disease, treatment and outcome data collected. | 6-9mth recruitment period, 18mth study duration.

SECONDARY OUTCOMES:
survival rates | 18 month period

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (59):
- Austria (4):
  - GSK Investigational Site, Graz
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Vienna
- Czechia (2):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Pilsen
- GSK Investigational Site, Tallinn, Estonia
- France (11):
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Draguignan
  - GSK Investigational Site, Lorient
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Perpignan
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Pierre-Bénite
  - GSK Investigational Site, Saint-Priest-en-Jarez
  - GSK Investigational Site, Strasbourg
- Germany (9):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Immenhausen, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Leer, Lower Saxony
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Hemer, North Rhine-Westphalia
  - GSK Investigational Site, Velbert, North Rhine-Westphalia
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Heraklion, Crete
  - GSK Investigational Site, Thessaloniki
- Hungary (2):
  - GSK Investigational Site, Mátraháza
  - GSK Investigational Site, Székesfehérvár
- Italy (5):
  - GSK Investigational Site, Lecce, Apulia
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Rozzano (MI), Lombardy
  - GSK Investigational Site, Orbassano (TO), Piedmont
  - GSK Investigational Site, Sassari, Sardinia
- Lithuania (3):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Klaipėda
  - GSK Investigational Site, Vilnius
- Netherlands (4):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Groningen
- Poland (6):
  - GSK Investigational Site, Gorzów Wielkopolski
  - GSK Investigational Site, Głuchołazy
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Warsaw
- Slovenia (2):
  - GSK Investigational Site, Golnik
  - GSK Investigational Site, Ljubljana
- South Korea (3):
  - GSK Investigational Site, Seongnam-si, Gyeonggi-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon, Gyeonggi-do
- Spain (4):
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Zaragoza